CLINICAL TRIAL: NCT06276088
Title: A Prospective Cohort Study of Plasma and Tissue SAA1 Levels in Cancer Patients to Predict Hyperprogression of Immunotherapy
Brief Title: Plasma and Tissue SAA1 Levels in Cancer Patients to Predict Hyperprogression of Immunotherapy
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2024-067
Record Dates: First submitted 2024-02-18; First posted 2024-02-23 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Immunotherapy; Hyperprogression; Biomarker
Keywords: SAA1; Immunotherapy; Hyperprogression; Pan-cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Tissue and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Immune checkpoint inhibitors have ushered in a new era of cancer treatment, bringing significant survival benefits to patients. However, some patients have accelerated tumor growth in the early stage of immunotherapy, called hyperprogression. The quality of life of patients with hyperprogression is seriously reduced, and there is no effective treatment at present, and the prognosis is extremely poor. Therefore, early identification of high-risk groups of hyperprogression is the key to prevent hyperprogression. However, there are no effective biomarkers to predict hyperprogression. By sequencing, proteomics and metabolomics analysis of clinical tissue and blood samples, we found that the level of SAA1 was significantly increased in patients with hyperprogression, and SAA1 was an effective marker for predicting hyperprogression in pan-cancer. We planned to conduct a multicenter, prospective cohort study to verify the reliability of SAA1 as a marker for predicting hyperprogression of immunotherapy in pan-cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years of age
2. Voluntarily sign informed consent
3. The pathological diagnosis was nasopharyngeal carcinoma, head and neck tumor, lung cancer, breast cancer, stomach cancer, colorectal cancer, glioma, esophageal cancer, liver cancer, bile duct cancer, cervical cancer, prostate cancer, bladder cancer and other malignant tumors
4. Need to be treated with immune checkpoint inhibitors
5. ECOG PS Score: 0/1.

Exclusion Criteria:

1. There are contraindications to immunotherapy
2. Combined with other tumors (basal cell or squamous cell skin cancer that has been cured, and cervical cancer in situ removed) External)
3. Patients had any serious coexisting medical conditions that could pose an unacceptable risk or negatively affect trial adherence. For example, unstable heart disease requiring treatment, chronic hepatitis, kidney disease, poor disease status, uncontrolled diabetes (fasting blood glucose > 1.5 × ULN), and mental illness.
4. At the investigator's discretion, those who was not considered to be suitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients who need to accept immunotherapy
Sampling Method: Probability Sample
Enrollment: 374 (Estimated)
Dates: Start 2024-02-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of hyperprogression | 2 years
  Incidence of hyperprogression will be calculated.

SECONDARY OUTCOMES:
Event-free survival | 3 years
  Event-free survival was defined as the time from the date of inclusion until hyperprogression or death from any cause.
Progression-free survival | 3 years
  Progression-free survival was defined as the time from the date of inclusion until disease progress or death from any cause.
Overall survival | 3 years
  Overall survival was defined as the time from the date of inclusion until death from any cause.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Nanfang hospital, Southern medical university, Guangzhou, Guangdong
  - Fujian Provinical Hospital, Fuzhou
  - Huizhou Central People's Hospital, Huizhou
  - Jieyang people's hospital, Jieyang
  - Meizhou People's Hospital, Meizhou Academy of Medical Sciences Meizhou, Meizhou

IPD SHARING:
Plan to Share IPD: No